CLINICAL TRIAL: NCT05576636
Title: The Effect of Simulation Education as an Approach to Patients With COVID-19 on Nursing Students' Perception and Fear of COVID-19 Disease: A Randomized Controlled Trial
Brief Title: COVID-19 Simulation Education on Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Nurten Terkes, Principal Investigator, Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MAKU-GO 2021/357
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: COVID-19 Pandemic; Simulation of Physical Illness
Keywords: nursing student; perception of illness; fear of death.
MeSH Terms: conditions — COVID-19; Necrophobia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Masking Description: They did not know if they were in the control and intervention group at the time of randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): After the pre-tests (the COVID-19 Disease Perception Scale, and the Fear of COVID-19 Scale) , the students were given simulation education for one months.
  Interventions: Behavioral: Simulation training
- Control Group (Experimental): The control group didn't apply any interference during the study. Participants in the control group continued their routine follow-up.
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: Simulation training — Expectations regarding the scenario were explained to the participants before the implementation. They were given information about the standard patient. Roles were distributed, and the implementation time of the scenario was announced. Written permission was obtained from students involved in the scenario. The intervention group was given scenario-based education appropriate for the approach to a standard patient with COVID-19. During the implementation of the scenario, the instructor did not interfere with students, and after the feedback, the "show-do" method was used to improve the incorrect skill steps. Two instructors evaluated students' performance on the standard patient simulation as "achieved-failed" and the application was recorded as a pre-test.
  Arms: Intervention group
Other: Control Group — The control group didn't apply any interference during the study. Participants in the control group continued their routine follow-up.
  Arms: Control Group

SUMMARY:
This study aims to determine the effect of simulation education as an approach to patients with COVID-19 on nursing students' perception and fear of the COVID-19 disease. This study was conducted in a randomized controlled trials with 86 nursing students from a university between November 10 and December 10, 2021.

ELIGIBILITY:
Inclusion Criteria:

* Nursing student and
* Agreeing to participate in the study

Exclusion Criteria:

* Refusing to participate in the study or quitting the study

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
Approach to COVID-19 Patient Form | 5 Minute
  This form was created by the researchers following a review of the literature (Collado-Boira et al., 2020; Cervera-Gasch, Gonz ́alez-Chorda ́, & Mena-Tudela, 2020; Kurt, & Dalkıran, 2021; Ulenaers, et al., 2021; Işık, Konuş, & Bakar, 2021) and was evaluated by 3 experts who had a PhD degree in the field, and necessary improvements were made in line with their suggestions. It consists of 14 items in total. This form includes interventions, such as "The mask should be worn before entering the patient room or care area" and "Disposable respiratory and face masks should be removed and discarded after leaving the patient's room or care area and closing the door." The correct application of these interventions was scored with "1 point" and the incorrect application with "0 points". Scores range between 0 and 14. As the scores increase, the accuracy level of the approach to the patient increases, as well.
The Fear of COVID-19 Scale | 5 Minute
  This scale was developed by Ahorsu et al. (2022), and its Turkish adaptation, validity, and reliability studies were performed by Ladikli et al. (2020). The scale has a single factor structure and consists of seven 5-point Likert-type (1 = strongly disagree; 5 = strongly agree) items. Scores on the scale range between 7 and 35. The higher the score is, the higher the fear of the COVID-19 pandemic is. Cronbach's alpha value of the scale is 0.82 (Ladikli et al., 2020).
The COVID-19 Disease Perception Scale | 5 Minute
  This scale was developed by Geniş et al. (2020). It consists of seven items. It has a five-point Likert-type structure and consists of two sub-dimensions. The total score is calculated by summing the scores of the items on the sub-dimension and dividing the results by the number of items on that sub-dimension. This operation yields a value between 1 and 5. High scores on the dangerousness sub-dimension indicate that the perceived dangerousness of the disease is high, and high scores on the contagiousness sub-dimension indicate that the perceived contagiousness of the disease is high. Cronbach's alpha value of the original scale is 0.78 (Geniş et al., 2020).

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Senturk, PhD, Study Chair — Burdur Mehmet Akif Ersoy University
Locations (1):
- Burdur Mehmet Akif Ersoy University, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All authors contributed to the interpretation, writing, and approval of the final manuscript.

REFERENCES:
- [Result] Hung CC, Kao HS, Liu HC, Liang HF, Chu TP, Lee BO. Effects of simulation-based learning on nursing students' perceived competence, self-efficacy, and learning satisfaction: A repeat measurement method. Nurse Educ Today. 2021 Feb;97:104725. doi: 10.1016/j.nedt.2020.104725. Epub 2020 Dec 16. PMID 33373813
- [Result] Huang CL. [Impact of Nurse Practitioners and Nursing Education on COVID-19 Pandemics: Innovative Strategies of Authentic Technology-Integrated Clinical Simulation]. Hu Li Za Zhi. 2021 Oct;68(5):4-6. doi: 10.6224/JN.202110_68(5).01. Chinese. PMID 34549401
- [Result] Almomani E, Sullivan J, Hajjieh M, Leighton K. Simulation-based education programme for upskilling non-critical care nurses for COVID-19 deployment. BMJ Simul Technol Enhanc Learn. 2020 Oct 21;7(5):319-322. doi: 10.1136/bmjstel-2020-000711. eCollection 2021. PMID 35515720